CLINICAL TRIAL: NCT06239584
Title: Generation of Lung Tumor Organoids From Patients Undergoing Diagnostic Bronchoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RS1766/22
Record Dates: First submitted 2024-01-12; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Generation of Lung Cancer Organoids
Keywords: Organoids.

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing diagnostic bronchoscopies for suspected lung cancer (Other): Preparation of organoids starting from lung tumor tissue collected during biopsies performed via diagnostic bronchoscopy according to standard clinical practice
  Interventions: Procedure: Biopsies performed via bronchoscopy

INTERVENTIONS:
Procedure: Biopsies performed via bronchoscopy — An additional amount of lung tumor tissue will be collected compared to that normally obtained as standard clinical practice, during bronchoscopy, al in order to increase the probability of successful generation of organoids

SUMMARY:
Interventional (low intervention level), non-pharmacological, prospective, feasibility pilot study of the preparation of organoids starting from lung tumor tissue collected during biopsies performed via diagnostic bronchoscopy according to standard clinical practice.

DETAILED DESCRIPTION:
Interventional, non-pharmacological, prospective, feasibility pilot study of the preparation of organoids starting from lung tumor tissue collected during biopsies performed via diagnostic bronchoscopy according to standard clinical practice. This protocol is classified as "interventional" (low intervention level) since that, if possible, an additional quantity of lung tumor tissue will be collected compared to that normally obtained as standard clinical practice, during bronchoscopy, al in order to increase the probability of successful generation of organoids. Involves the prospective recruitment of patients undergoing diagnostic bronchoscopies for suspected lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected diagnosis of centrally located and accessible lung cancer endoscopically;
* patients for whom it is indicated to undergo in-depth diagnostic testing through bronchoscopy for the purpose of determining the histotype of the lung neoplasm, according to clinical practice standard;
* aged over 18;
* patients who express informed consent to the study.

Exclusion Criteria:

* medical contraindication to taking biopsy samples;
* medical contraindication to carrying out endoscopic investigations;
* patients with suspected lung cancer not accessible endoscopically;
* patients with lung neoformation already subjected to diagnostic sampling;
* contraindications to taking an additional quantity of tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-02-02 (Estimated)

PRIMARY OUTCOMES:
Preparation of at least 10 tumor organoid cultures lung | 12 months
  Preparation of at least 10 tumor organoid cultures lung derived from patients undergoing diagnostic bronchoscopy. This study will allow define the success rate in the generation of organoids from diagnostic bronchoscopies.
  Performing a diagnostic bronchoscopy (scheduled as per clinical practice).

SECONDARY OUTCOMES:
Correspondence between the generated organoids and the tissue tumor of origin | 12 months
  Verify the correspondence between the generated organoids and the tissue tumor of origin. Expecting to carry out broad-spectrum molecular investigations, such as DNA mutational analysis via Whole Exome Sequencing (WES), and expression profiling gene through RNA-sequencing (RNAseq),through the use of the AllPrep DNA/RNA/miRNA Universal Kit (Quiagen) and of the tumors of origin taken through bronchoscopy diagnostics, as well as derived organoid cultures (PDO).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Blandino, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy